CLINICAL TRIAL: NCT03548155
Title: Berberine Effects on Clinical Symptoms and Metabolic Disturbance as an Adjunctive Therapy in Patients With Schizophrenia: a Randomized Double-blind Placebo-controlled Study
Brief Title: Berberine Effects on Clinical Symptoms and Metabolic Disturbance in Patients With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Anding Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BBR-SCH-2015
Record Dates: First submitted 2018-05-14; First posted 2018-06-07 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2018-05

CONDITIONS: Schizophrenia; Therapeutics
Keywords: schizophrenia；berberine；symptoms；inflammation
MeSH Terms: conditions — Schizophrenia | interventions — Berberine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- berberine group (Experimental)
  Interventions: Drug: Berberine; Drug: atypical antipsychotic
- control group (Placebo Comparator)
  Interventions: Drug: atypical antipsychotic; Drug: placebo

INTERVENTIONS:
Drug: Berberine — Berberine 300mg（three times a day） plus any atypical antipsychotic drug
  Arms: berberine group
Drug: atypical antipsychotic — Any atypical antipsychotic drug as the basic treatment
Drug: placebo — The placebo were matched to Berberine in shape, smell and colour and capsules were sealed in identical bottles
  Arms: control group

SUMMARY:
The study was a 8-week, randomized, double-blind, placebo-controlled trial. Berberine (300 mg，three times a day), as an adjuvant therapy has been used on the basis of the Second-generation antipsychotics（SGAs） monotherapy. All participants were randomly divided into two groups.Any SGA + berberine (BBR) or any SGA +placebo.Positive and Negative Syndrome Scale (PANSS) has been used for psychiatric symptoms.The treatment Emergent Symptom Scale(TESS) has been used for evaluate adverse effects.Glucose and lipid profile, inflammatory factors，adiponectin，leptin were obtained at 0, 4,8 weeks.

DETAILED DESCRIPTION:
Glucose and lipid profile:Fasting blood samples for Fasting blood glucose(FBG),Insulin, Hemoglobin A1c(HbA1c), Total cholesterol(TC), Low-density lipoprotein cholesterol(LDL-C),High-density lipoprotein cholesterol(HDL-C), Triglycerides (TG),Apolipoprotein A(ApoA),Apolipoprotein B(ApoB),Lipoprotein-a(Lp-a) .

Inflammatory factors:C-reaction protein(CRP),Interleukine-1 beta(IL-1β), Interleukine-6 (IL-6), Tumor necrosis factor-α (TNF-α).

ELIGIBILITY:
Inclusion Criteria:

* Individuals who aged 18 to 65 years
* Meet the diagnosis of schizophrenia according to DSM-IV
* Monotherapy of atypical antipsychotics for 4 weeks or more
* At least 60 for Positive and Negative Syndrome Scale (PANSS)
* Female subjects will be eligible to participate in the study if they are of non-childbearing potential or of child-bearing potential
* Sign the informed consent form

Exclusion Criteria:

* Individuals who with diagnosis of other psychiatric disorders except schizophrenia according to DSM-IV
* Refused to provide informed consent
* Significant medical illnesses including uncontrolled hypertension, diabetes, seizure disorder, severe cardiovascular, cerebrovascular, pulmonary, or thyroid diseases
* Currently on anti-inflammatory or immunosuppressant medication including oral steroids and history of chronic infection (including tuberculosis, HIV and hepatitis), malignancy, organ transplantation, blood dyscrasia, central nervous system demyelinating disorder, and any other known autoimmune or inflammatory condition.

Ages: 18 Years to 62 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2014-07-24 (Actual); Primary Completion 2015-12-14 (Actual); Study Completion 2017-05-08 (Actual)

PRIMARY OUTCOMES:
Changes of negative symptoms | changes within 0,4,8weeks
  Positive and Negative Syndrome Scale（PANSS）has been used to assess symptom severity in schizophrenia.Of the items included in PANSS ,seven constitute a Positive scale,seven form a Negative scale and sixteen constitute a General Psychopathology scale.7-point rating instrument was conceived.A total Score is computed three subscales.Minimum scores is 30 and maximum scores is 210.The higher score are considered the psychiatric symptoms more serious.

SECONDARY OUTCOMES:
Changes of Fasting blood samples for Fasting blood glucose(FBG) | changes within 0,4,8 weeks
  The levels of FBG has been obtained at 3 point intervals: 0, 4, 8 weeks
Changes of Insulin | changes within 0,4,8 weeks
  The levels of Insulin has been obtained at 3 point intervals: 0, 4, 8 weeks
Changes of TC | changes within 0,4,8 weeks
  The levels of TC has been obtained at 3 point intervals: 0, 4, 8 weeks
Changes of TG | changes within 0,4,8weeks
  The levels of TG has been obtained at 3 point intervals: 0, 4, 8 weeks
Changes of HDL-C | changes within 0,4,8weeks
  The levels of HDL-C has been obtained at 3 point intervals: 0, 4, 8 weeks
Changes of LDL-C | changes within 0,4,8weeks
  The levels of LDL-C has been obtained at 3 point intervals: 0, 4, 8 weeks
Safety | changes within 0,4,8weeks
  Evaluate the safety of berberine
Changes of CRP | changes within 0,4,8weeks
  The levels of CRP has been obtained at 3 point intervals: 0, 4, 8 weeks
Changes of IL-1β | changes within 0,4,8weeks
  The levels of IL-1β has been obtained at 3 point intervals: 0, 4, 8 weeks
Changes of IL-6 | changes within 0,4,8weeks
  The levels of IL-6 has been obtained at 3 point intervals: 0, 4, 8 weeks
Changes of TNF-α | changes within 0,4,8weeks
  The levels of TNF-α has been obtained at 3 point intervals: 0, 4, 8 weeks

REFERENCES:
- [Derived] Li M, Qiu Y, Zhang J, Zhang Y, Liu Y, Zhao Y, Jia Q, Fan X, Li J. Improvement of adjunctive berberine treatment on negative symptoms in patients with schizophrenia. Eur Arch Psychiatry Clin Neurosci. 2022 Jun;272(4):633-642. doi: 10.1007/s00406-021-01359-4. Epub 2022 Jan 17. PMID 35037116